CLINICAL TRIAL: NCT04960475
Title: An Observational Study of the Relationship Between Negative Emotion, Fear-Avoidance Belief and Quality of Life in Patients With Chronic Ankle Sprain
Brief Title: Study of Negative Emotion, Fear-Avoidance Belief and Quality of Life in Patients With Ankle Sprain
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021078
Record Dates: First submitted 2021-07-04; First posted 2021-07-13 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-07

CONDITIONS: Chronic Ankle Sprain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A/D group: Chronic ankle sprain patient with anxity or depression
  Interventions: Other: Hospital Anxious and Depression(HADS); Other: Fear-Avoidance Belief Questionnaire (FABQ); Other: The MOS 36-Item Short From Health Survey (SF-36)
- Control group: Chronic ankle sprain patient with no emotional issues
  Interventions: Other: Hospital Anxious and Depression(HADS); Other: Fear-Avoidance Belief Questionnaire (FABQ); Other: The MOS 36-Item Short From Health Survey (SF-36)

INTERVENTIONS:
Other: Hospital Anxious and Depression(HADS) — The assessment content in the scale is divided into two parts: anxiety and depression. Anxiety is an unexplained state of restlessness, manifested as tension, fear, and panic all day long. Depression is manifested as depression, slow thinking, decreased volition and physical symptoms. The two parts are scored separately. A total score of 0-7 means normal, a total score of 8-10 means mild depression/anxiety, a total score of 11-14 means moderate depression/anxiety, and a total score of 15-21 means severe depression/ anxiety.
Other: Fear-Avoidance Belief Questionnaire (FABQ) — FABQ is a self-assessment questionnaire with 16 options. Each option has 7 levels of 0-6 points, representing totally disagree, uncertain, and totally agree; there are 2 subscales, and one subscale measures the fear-avoidance in physical activity, another subscale measures fear-avoidance of work. The final score of FABQ is the superposition of the value of each item. A high score indicates a high level of fear-avoidance beliefs.
Other: The MOS 36-Item Short From Health Survey (SF-36) — The SF-36 is a multi-purpose survey designed to capture adult patients' perceptions of their own health and well-being. The SF-36 has 36 items grouped in 8 dimensions: physical functoning, physicial and emotional limitations, social functioning, bodily pain, general and mental health.

SUMMARY:
This study intends to investigate the negative emotions, fear-avoidance beliefs, and quality of life in patients with chronic ankle sprains to explore the relationship between negative emotions such as anxiety and depression, fear-avoidance beliefs, and their impact on quality of life.

DETAILED DESCRIPTION:
Research design: This study is an observational study. It is planned to recruit a total of 120 patients with ankle sprain injury who meet the selection criteria from the Rehabilitation Department of Peking University Third Hospital. They will be divided into an anxiety and depression group and a control group based on anxiety and depression scale. Basic information, anxiety and depression scales, fear-avoidance beliefs score and quality of life score of two groups will be compared and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Ankle sports injury time> 6 months;
* age 18-50 years;
* no pain in daily activities, or a numerical rating scale (NRS) 6 points or less;
* no mechanical instability of the ankle joint and obvious restriction in joint movement ;
* agree to participate in this study.

Exclusion Criteria:

* acute inflammation of lower limb joints;
* new or unhealed lower limb fractures;
* history of lower limb surgery within 3 months;
* lower limb pain caused by other diseases (such as lumbar disease, vascular disease, etc.);
* speech and cognitive impairment
* other diseases that cannot participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ankle sprains are the most common injury in everyday life, military training and sports. Forty percent of people with ankle sprains develop chronic ankle instability, including mechanical ankle instability and functional ankle instability. Mechanical ankle instability is usually caused by structural changes in the ligamentous tissue around the ankle, kinematic damage, synovial changes or degenerative joint disease. Functional ankle instability refers to the subjective perception of instability during daily life or sports. Most patients do not require surgery, and clinical examination reveals only minor swelling and localized pressure pain, but rarely severe structural damage to the joint with limited range of motion and joint instability. However, many patients with chronic functional instability of the ankle joint due to ankle sprain are unable to resume normal work and life due to emotional anxiety and repeatedly seek medical attention.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
FABQ score | 1 hr
  the total score of Fear-Avoidance Belief Questionnaire
SF-36 score | 1 hr
  the score of SF36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hongying Zhong, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No